CLINICAL TRIAL: NCT06785870
Title: Evaluation of Erythrocytosis Prospective Cohort Study (EVEREST): Diagnosis, Management and Longitudinal Outcomes in Patients with Elevated Hemoglobin
Brief Title: EVAluation of Erythrocytosis PRospEctive Cohort STudy
Acronym: EVEREST
Status: Not yet recruiting | Type: Observational
Sponsor: Cyrus Hsia (Other)
Responsible Party: Sponsor-Investigator, Cyrus Hsia, Hematologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: HSREB125939
Record Dates: First submitted 2024-09-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Erythrocytosis; Polycythemia; Polycythemia Secondary; Polycythemia Vera; Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Polycythemia Vera (PV); Polycythemia; Familial; Polycythemia, Primary
Keywords: Prospective; Observational Study; Erythrocytosis; Polycythemia; Patient Registry; Diagnosis; Management; Outcomes
MeSH Terms: conditions — Polycythemia; Polycythemia Vera; Polycythemia, primary familial and congenital; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Erythrocytosis patients: Adult patients (>=18 years) referred to hematology clinics at London Health Sciences Centre (LHSC) with erythrocytosis or polycythemia with hemoglobin levels >=165 g/L in males or >=160 g/L in females at the time of initial clinic visit.

SUMMARY:
The EValuation of ERythrocytosis pRospEctive cohort STudy (EVEREST) is a prospective study designed to shed light on these key questions in the diagnosis, management, and clinical outcomes in patients with elevated hemoglobin (erythrocytosis). This longitudinal, prospective study will generate high quality data that can help inform the optimal approach to diagnosis and management in this patient population.

DETAILED DESCRIPTION:
The EVAluation of Erythrocytosis pRospEctive cohort STudy (EVEREST) is a prospective, longitudinal, observational study designed to provide insights into the diagnosis, management, and outcomes of patients with elevated hemoglobin (erythrocytosis). This study aims to address key gaps in understanding the underlying causes, diagnostic approaches, and clinical outcomes of patients presenting with erythrocytosis in real-world clinical settings.

Erythrocytosis, defined as an elevated hemoglobin concentration, is a frequent reason for referral to hematology and presents substantial diagnostic and therapeutic challenges. The condition may arise from primary causes, such as polycythemia vera (PV), or secondary causes, including chronic hypoxia, erythropoietin-secreting tumors, medications, and exogenous testosterone use. Despite advances in diagnostic tools, there remains considerable uncertainty about the most effective ways to evaluate and manage erythrocytosis, particularly in distinguishing secondary from primary causes and in mitigating associated risks such as arterial and venous thrombosis.

EVEREST is designed to address these knowledge gaps by enrolling a diverse cohort of patients referred to hematology for evaluation of erythrocytosis. Participants will undergo comprehensive clinical evaluation and assessment of potential underlying causes. Data will be collected longitudinally to evaluate real-world management practices, such as the use of phlebotomy, cytoreductive therapy, and antithrombotic agents, and to document clinical outcomes, including rates of thrombosis, bleeding, disease progression, and mortality.

The study has four main objectives:

1. To prospectively measure the incidence of various causes of erythrocytosis in patients referred for elevated hemoglobin levels.
2. To prospectively evaluate the diagnostic accuracy of the JAKPOT prediction rule, a simple prediction rule using complete blood count parameters, for identifying JAK2-positive erythrocytosis/polycythemia vera and differentiating it from secondary causes.
3. To evaluate real-world management strategies for patients with erythrocytosis.
4. To document longitudinal clinical outcomes, including thrombosis, bleeding, disease progression, and survival.

EVEREST aims to recruit 1,500 adult patients across participating clinics. Participants will be followed for clinical outcomes, and data will be collected to better characterize therapeutic approaches utilized in routine clinical care. This study seeks to generate evidence that will inform clinical practice and improve patient care for patients with erythrocytosis.

Outcome Measures EVEREST is a prospective observational study which will investigate multiple interrelated aspects of erythrocytosis, encompassing its causes, diagnostic evaluation, management strategies, and clinical outcomes. Two co-primary outcome measures have been selected to reflect the study's main objectives to measure the incidence and causes of erythrocytosis and the diagnostic accuracy of the JAKPOT prediction rule. Additionally, secondary outcome measures will focus on real-world management strategies and longitudinal clinical outcomes, providing further insights to inform patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>=18 years) referred to hematology clinics at London Health Sciences Centre with hemoglobin levels >=165 g/L in males or >=160 g/L in females.
2. Patients capable of providing informed consent.
3. Age >= 18 years.

Exclusion Criteria:

1. Patients <18 years.
2. Patients without erythrocytosis.
3. Patients incapable of providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EVEREST will recruit adult patients evaluated for erythrocytosis, hemoglobin levels >=165 g/L in males or >=160 g/L in females, in hematology clinics at London Health Sciences Centre.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Causes of Erythrocytosis | 5 years
  The study will measure the incidence of primary and secondary causes of erythrocytosis, including polycythemia vera (PV), chronic hypoxia, medication use (e.g., SGLT2 inhibitors, testosterone), and other secondary causes. Data will be derived from clinical records and diagnostic investigations conducted as part of routine care.
  Unit of Measure: Proportion of participants (%) and count (n) categorized by cause over the study duration.
Diagnostic Accuracy of the JAKPOT Prediction Rule | 5 years
  The diagnostic accuracy of the JAKPOT prediction rule will be assessed for differentiating JAK2-positive erythrocytosis/PV from other causes. Measures will include sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).
  Unit of Measure: Sensitivity (%), specificity (%), PPV (%), and NPV (%).

SECONDARY OUTCOMES:
Frequency of Management Strategies | 5 years
  The study will document the proportion of participants receiving various management strategies, including phlebotomy, cytoreductive therapy, antiplatelet agents (e.g., aspirin), and anticoagulants. Data will include timing, frequency, and type of intervention, as recorded in clinical records.
  Unit of Measure: Proportion of participants (%) and count (n) receiving each management strategy.
Incidence of Thrombotic Events | 5 years
  Thrombotic events, including venous thromboembolism (deep vein thrombosis, pulmonary embolism) and arterial thrombosis (ischemic stroke, myocardial infarction), will be documented based on clinical records and imaging results. Standard definitions will be applied for classification.
  Unit of Measure: Events per 100 person-years.
Incidence of Bleeding Events | 5 years
  Bleeding events, categorized as major or clinically relevant non-major bleeding following ISTH definitions, will be measured. Data will include site, severity, and clinical consequences of bleeding.
  Unit of Measure: Events per 100 person-years.
Disease Progression | 5 years
  Disease progression, defined as transformation to myeloproliferative neoplasms (e.g., myelofibrosis, myelodysplastic syndrome, acute leukemia) or other hematologic malignancies, will be captured. Progression will be classified using WHO criteria and supported by clinical and laboratory data.
  Unit of Measure: Incidence per 100 person-years.
Mortality | 5 years
  Mortality data will include all-cause and cause-specific deaths, categorized as cardiovascular-related, thrombotic, hemorrhagic, or due to disease progression. Cause-specific data will be confirmed by clinical documentation or autopsy reports where available.
  Unit of Measure: Incidence per 100 person-years.

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided